CLINICAL TRIAL: NCT00782730
Title: Assessment of Third Trimester Post-void Residual Along With Determining Validity of the Bladder Scanner in the Third Trimester of Pregnancy and Postpartum
Brief Title: Assessment of Third Trimester Post-void Residual and Validation of Bladder Scanner in Pregnancy and Post-partum
Status: Completed | Type: Observational
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Michael Stitely, Adjunct Associate Professor, West Virginia University
Other Study IDs: H-20862
Record Dates: First submitted 2008-10-29; First posted 2008-10-31 (Estimated); Last update posted 2013-06-13 (Estimated); Status verified 2013-06

CONDITIONS: Pregnancy
Keywords: bladder volume measurement; pregnancy; bladder function; Postvoid residual volume assessment; Bladder volumes

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bladder Scan Group: Patients who agree to enroll in the trial and allow their known bladder volumes and residual bladder volumes to be measured by actual volumes retrograde instilled, and also by bladder scanner ultrasound.

SUMMARY:
This will be a descriptive study measuring the post-void residual of patients in the third trimester and postpartum. Also, bladder scan values will be compared to the amount of urine obtained from a Foley catheter to determine the accuracy of the bladder scanner in the third trimester and postpartum.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years.
* Having a non-emergent Cesarean Delivery or labor epidural placed.

Exclusion Criteria:

* Age less than 18 years.
* Emergent Cesarean delivery.
* No epidural labor analgesia.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients undergoing elective or non-emergent Cesarean delivery will be asked to enroll. Also adult patients having a labor epidural placed during labor will be asked to participate.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2008-10; Primary Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Define normal post-void residual volume in third trimester pregnancy and post-partum. | 12-24 hours

SECONDARY OUTCOMES:
Calculate the validity of measurements form the bladder scanner ultrasound for bladder volumes during the third trimester of pregnancy and post-partum. | 12-24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Stitely, MD, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University, Morgantown, West Virginia, United States